CLINICAL TRIAL: NCT04292912
Title: Phase I, Open-Label, Multi-Center Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of GSK2798745 After 28 Day Repeat Oral Administration to Adults With Diabetic Macular Edema
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK2798745 in Participants With Diabetic Macular Edema
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated as the study met the prespecified threshold for futility of less than (<) 20 percentage (%), based on interim analysis (IA).
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212669
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-08

CONDITIONS: Macular Edema
Keywords: Diabetic macular edema; GSK2798745; Refraction; Visual acuity.
MeSH Terms: conditions — Macular Edema | interventions — GSK2798745

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, single arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GSK2798745 (Experimental): Eligible participants received single dose of GSK2798745 for 28 days. Participants were instructed to have GSK2798745 about the same time each day.
  Interventions: Drug: GSK2798745

INTERVENTIONS:
Drug: GSK2798745 — GSK2798745 will be administered.

SUMMARY:
The study will be composed of 3 periods for all participants: Screening, 28-day Treatment period, and Follow-up visit (approximately 28 days after the final dose).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 to 75 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of diabetes mellitus (type 1 or type 2).
* Confirmation of DME with center involvement in at least one eye by fluorescein angiography.
* Confirmation of retinal thickening (diabetic macular edema) involving the center of the fovea in the study by Investigator.
* Best Corrected Visual Acuity (BCVA) letter score of 80 letter or worse (Snellen equivalent: equivalent to 20/25) or worse in the study eye.
* Safe to withhold treatment of the study eye with laser photocoagulation, intravitreal steroid injection, or intravitreal vascular endothelial growth factor (VEGF) inhibitor for the duration of the study.
* Body weight greater than equal to (>=) 50 kilograms (kg) and Body mass index (BMI) within the range 18 to 43 kg per square meter (inclusive) at screening.
* Male participants must agree to refrain from donating sperm, plus either be abstinent from heterosexual or homosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or must agree to use acceptable contraception/barrier to use acceptable contraceptive methods if their partner is of childbearing potential. This criterion must be followed from the first dose of study treatment until the follow-up visit.
* A female participant is eligible to participate if she is not of childbearing potential.

Exclusion Criteria:

* Additional eye disease in the study eye that in the opinion of the Investigator could compromise assessment.
* History of choroidal neovascularization in the study eye, or current choroidal neovascularization in the fellow eye requiring treatment.
* Active Proliferative diabetic retinopathy (PDR) in the study eye or untreated active PDR in the fellow eye.
* Ischemic maculopathy on fluorescein angiography.
* Intraocular surgery or laser photocoagulation in the study eye within 90 day.
* Use of intravitreal ranibizumab,or bevacizumab within 42 days (6 weeks), or aflibercept within 56 days (8 weeks) of dosing in the study eye.
* Use of intraocular steroids in the study eye within 180 days of dosing.
* Use of or expected need for intravitreal or intraocular treatment in the study eye during course of the study.
* Use of any systemically administered anti-angiogenic agent within 6 months of dosing.
* Evidence of vitreomacular traction as determined by the Investigator.
* Uncontrolled intraocular pressure in the study eye despite treatment with glaucoma medication.
* Within 6 months prior to the Screening Visit, use of medications known to be toxic to the retina, lens or optic nerve
* Uncontrolled diabetes as indicated by glycated hemoglobin (HbA1c) >12% at Screening.
* Active ulcer disease or gastrointestinal bleeding by history within 6 months of screening or by exam at the time of screening.
* Certain type of liver disease.
* Participant who, in the Investigator's opinion, poses a significant suicide risk.
* History or current evidence of any serious or clinically significant cardiac, gastrointestinal, renal, endocrine, neurologic, hematologic, infectious or other condition that is uncontrolled.
* Corrected (QTc) interval >450 milliseconds (msec) or QTc >480 msec in participants with bundle branch block.
* Use of certain medications that may interfere with the study medication or eye assessments (these will be identified by the study doctor).
* Current enrollment, or recent participation in a study of investigational intervention or medical research.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation in the study.
* Any other reason the investigator deems the participant should not participate in the study.
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (6):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Winter Haven, Florida
  - GSK Investigational Site, Shirley, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, McAllen, Texas
- Australia (4):
  - GSK Investigational Site, Castle Hill, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Melbourne, Victoria
- GSK Investigational Site, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants who passed screening and eligible for the study with intention to dose were enrolled in the study. A total of 16 participants were included who received at least one dose of study treatment for 28 days. Of which, 9 completed the study and 7 participants discontinued the study. The study was terminated early due to meeting the interim futility.
Pre-assignment Details: The analysis population included 16 participants who received at least 1 dose of study treatment. This included 6 participants from prematurely closed site due to protocol violations.
Period: Overall Study
Arm/Group | GSK2798745
Started | 16
Completed | 9
Not Completed | 7
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Arm/Group | GSK2798745
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 4
  White | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abnormal Ophthalmic Examination Findings
Description: Ophthalmic examinations for Pupil motility and confrontation visual field examination, slit lamp evaluation of anterior ocular structures, intraocular pressure measurement and optical coherence tomography (OCT) was performed on left and right eye. Participants with data including abnormalities of potential clinical importance is listed here.
Time Frame: Up to Day 28
Population: Modified safety population comprised of all participants who received at least one dose of study treatment. Only those participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2798745
Number analyzed (Participants) | 10
Participants
  Eyelids and Lashes | 0
  Pupil motility | 0
  Confrontation visual field examination | 0
  Slit lamp evaluation of anterior ocular structures | 0
  Intraocular pressure measurement, Left eye: number analyzed (Participants) | 9
  Intraocular pressure measurement, Left eye | 1
  Intraocular pressure measurement, Right eye: number analyzed (Participants) | 9
  Intraocular pressure measurement, Right eye | 1
  OCT center subfield, Left eye | 0
  OCT center subfield, Right eye | 1

2. Primary Outcome: Mean Change From Baseline to Day 28 in Visual Acuity
Description: Best-correct visual acuity (BCVA) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts. The visual function of the study eye was assessed using the ETDRS protocol. ETDRS letters score can be calculated when 20 or more letters are read correctly at 4.0 meters (m); the visual acuity letter score is equal to the total number of letters read correctly at 4.0 m plus 30. If less than 20 letters are read correctly at 4.0 m, the visual acuity letter score is equal to the total number of letters read correctly at 4.0 m (number of letters recorded on line 1.0), plus the total number of letters read correctly at 1.0 m in the first six lines. The score ranges from 0-100 where a higher score represents better visual functioning. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: Pharmacodynamics (PD) analysis set included all participants from the modified Safety population who had at least 1 post-baseline non-missing PD assessment.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
Letters | 1.6 (4.67)

3. Primary Outcome: Mean Change From Baseline to Day 28 in Body Weight
Description: Physical examination included the measuring of body weight and evaluated at indicated time points. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
kilogram (kg) | -0.34 (1.157)

4. Primary Outcome: Mean Change From Baseline to Day 28 in Body Temperature
Description: Physical examination included the measuring of body temperature and evaluated at indicated time points. The change from Baseline was calculated by subtracting Baseline value from post-Baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degree Celsius (°C)
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
Degree Celsius (°C) | 0.04 (0.416)

5. Primary Outcome: Mean Change From Baseline to Day 28 in Vital Signs for Systolic Blood Pressure and Diastolic Blood Pressure
Description: The change from baseline for Systolic Blood Pressure (SBP) and Diastolic blood Pressure (DBP) was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
mmHg
  SBP on Day 28 | 5.67 (13.611)
  DBP on Day 28 | 1.44 (9.167)

6. Primary Outcome: Mean Change From Baseline to Day 28 in Pulse Rate
Description: Pulse rate was measured at indicated time points. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beats per Minute (beats/min)
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
Beats per Minute (beats/min) | -1.33 (10.368)

7. Primary Outcome: Mean Change From Baseline to Day 28 in 12-lead Electrocardiogram (ECG) Findings
Description: The 12-lead ECGs was obtained at indicated timepoints during the study. The standard ECG criteria of potential clinical importance were 1) absolute QTc Interval, > 450 milliseconds (msec), 2) absolute PR Interval, <110 msec, 3) absolute QRS Interval, < 75 msec and 4) increase from baseline in QTc > 60 msec. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: The intensive pharmacokinetics (PK) analysis population included all participants from the modified Safety population who had intensive PK sampling on Day 7 and Day 28. However, since only one participant consented to intensive PK and this participant withdrew early, before Day 28, data for this endpoint were not collected.
Arm/Group | GSK2798745
Number analyzed (Participants) | 0

8. Primary Outcome: Mean Change From Baseline to Day 28 in Alanine Amino Transferase (ALT), Alkaline Phosphatase (AP), Aspartate Amino Transferase (AST), and Creatine Kinase
Description: Summary of changes from baseline in laboratory parameters were assessed. The analysis included liver function tests for ALT, AP, AST, Creatine kinase and evaluated at indicated time points. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Microkatal per Litre (ukat/L)
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
Microkatal per Litre (ukat/L)
  Alanine Aminotransferase (ALT) | -0.01 (0.087)
  Alkaline Phosphatase | -0.11 (0.179)
  Aspartate Aminotransferase | -0.02 (0.134)
  Creatine Kinase | 0.10 (0.318)

9. Primary Outcome: Mean Change From Baseline to Day 28 in Calcium, Glucose, Potassium, Sodium, and Urea Nitrogen
Description: Summary of changes from baseline in clinical chemistry parameters. The parameters included were calcium, glucose, potassium, sodium and urea nitrogen and evaluated at indicated time points. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
Millimoles per Liter (mmol/L)
  Calcium | 0.0 (0.107)
  Glucose | 2.15 (3.485)
  Potassium | 0.04 (0.354)
  Sodium | 1.33 (2.550)
  Urea Nitrogen | -0.46 (2.606)

10. Primary Outcome: Mean Change From Baseline to Day 28 in Creatinine, Total Bilirubin, and Direct Bilirubin
Description: Summary of changes from baseline in clinical chemistry parameters. The parameters analyzed were creatinine, total bilirubin and direct bilirubin and evaluated at indicated timepoints. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (umol/L)
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
Micromoles per Liter (umol/L)
  Creatinine | 1.18 (10.237)
  Total Bilirubin | 0.92 (3.923)
  Direct Bilirubin | 0.52 (0.995)

11. Primary Outcome: Mean Change From Baseline to Day 28 in Clinical Chemistry Parameter Values of Protein
Description: Summary of changes from baseline in clinical chemistry parameter, Protein. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
Grams per Liter (g/L) | -0.89 (4.014)

12. Primary Outcome: Mean Change From Baseline to Day 28 in Clinical Chemistry Parameter Values of Cardiac Troponin
Description: Summary of changes from baseline in clinical chemistry parameters for Cardiac troponin. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
nanograms per milliliter (ng/mL) | 0.00 (0.004)

13. Primary Outcome: Mean Change From Baseline to Day 28 in Basophils, Eosinophils, Leukocytes, Monocytes, Lymphocytes, Neutrophils, and Platelets
Description: Summary of changes from baseline in hematology. The parameters analyzed were Basophils, Eosinophils, Leukocytes, Monocytes, Lymphocytes, Neutrophils and Platelets at indicated time points. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter
Arm/Group | GSK2798745
Number analyzed (Participants) | 8
Giga (10^9) cells per liter
  Basophils | 0.00 (0.014)
  Eosinophils | 0.02 (0.092)
  Leukocytes | 0.19 (1.860)
  Lymphocytes | -0.13 (0.506)
  Monocytes | -0.02 (0.106)
  Neutrophils | 0.34 (1.450)
  Platelets | -0.50 (23.952)

14. Primary Outcome: Mean Change From Baseline to Day 28 in Mean Corpuscular Hemoglobin Concentration (MCHC) and Hemoglobin (Hb)
Description: Summary of changes from baseline in hematology. The parameters analyzed were MCHC and Hb at indicated time points. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | GSK2798745
Number analyzed (Participants) | 8
g/L
  MCHC | -1.63 (9.709)
  Hb | -0.88 (5.693)

15. Primary Outcome: Mean Change From Baseline to Day 28 in Mean Corpuscular Hemoglobin
Description: Summary of changes from baseline in mean corpuscular hemoglobin at indicated time points. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Picograms per cell (pg/cell)
Arm/Group | GSK2798745
Number analyzed (Participants) | 8
Picograms per cell (pg/cell) | -0.44 (0.703)

16. Primary Outcome: Mean Change From Baseline to Day 28 in Mean Corpuscular Volume (MCV)
Description: Summary of changes from baseline in hematology MCV assessment. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | GSK2798745
Number analyzed (Participants) | 8
Femtoliter | -1.10 (2.943)

17. Primary Outcome: Mean Change From Baseline to Day 28 in Erythrocytes
Description: Summary of changes from baseline in erythrocytes at indicated time points. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter
Arm/Group | GSK2798745
Number analyzed (Participants) | 8
10^12 cells per Liter | 0.04 (0.213)

18. Primary Outcome: Mean Change From Baseline to Day 28 in Hematocrit
Description: Summary of changes from baseline in hematocrit parameter at indicated time points. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | GSK2798745
Number analyzed (Participants) | 8
Proportion of red blood cells in blood | 0.0 (0.018)

19. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Ocular and Non-ocular AEs and SAEs
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury. Data has been presented for number of participants with ocular and non-ocular AEs and SAEs.
Time Frame: Until follow-up (Up to Day 56)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2798745
Number analyzed (Participants) | 16
Participants
  AEs | 4
  SAEs | 0
  Ocular AEs | 2
  Ocular SAEs | 0
  Non-ocular AEs | 3
  Non-ocular SAEs | 0

20. Primary Outcome: Mean Change From Baseline to Day 28 in Center Subfield Retinal Thickness as Measured by Spectral-Domain Optical Coherence Tomography (SD-OCT)
Description: The SD-OCT effect is a pharmacodynamics (PD) measure of daily repeated dosing of GSK2798745. The mean change from baseline in macular thickness was measured by SD-OCT in the study eye after 28 days of dosing. Measurements was obtained by an appropriately trained photographer/technician using SD-OCT equipment that has been approved by a central reader. The change from baseline was calculated by subtracting baseline value from post-baseline value.
Time Frame: Baseline and Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrometer (um)
Arm/Group | GSK2798745
Number analyzed (Participants) | 9
Micrometer (um) | -3.6 (35.05)

21. Secondary Outcome: Plasma Concentrations of GSK2798745
Description: Blood samples were collected at indicated time points for plasma concentrations of GSK2798745.
Time Frame: Day 7 (Pre-dose, 0.5 hour [h], 1h, 2h, 3h, 4h, 6h, 8h) and Day 28 (Pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h)
Population: The pharmacokinetic population included all participants from the modified safety population who received at least one dose of study treatment for whom PK sample was obtained and analyzed. Only those participants with evaluable PK data at the specified time points were used for analysis. Overall number of participants analyzed=number of participants contributed to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | GSK2798745
Number analyzed (Participants) | 5
nanograms per milliliter
  Day 7 | 6.24 (70.4)
  Day 28: number analyzed (Participants) | 3
  Day 28 | 8.61 (125.1)

22. Secondary Outcome: Plasma Concentrations of Major Metabolite M1
Description: Blood samples were collected at indicated time points for PK analysis of major metabolite of GSK2798745.
Time Frame: Day 7 (Pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h) and Day 28 (Pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | GSK2798745
Number analyzed (Participants) | 5
nanograms per milliliter
  Day 7 | 9.32 (49.9)
  Day 28: number analyzed (Participants) | 3
  Day 28 | 9.83 (64.8)

23. Secondary Outcome: Absorption Rate of GSK2798745
Description: Blood samples were collected at indicated time points for PK analysis of GSK2798745 absorption rate.
Time Frame: Day 28
Population: The intensive PK analysis population included all participants from the modified Safety population who had intensive PK sampling on Day 7 and Day 28. However, since only one participant consented to intensive PK and this participant withdrew early, before Day 28, data for this endpoint were not collected.
Arm/Group | GSK2798745
Number analyzed (Participants) | 0

24. Secondary Outcome: Clearance of GSK2798745
Description: Blood samples were collected at indicated time points for PK parameters including clearance of GSK2798745.
Time Frame: At Day 28
Population: as for outcome 23
Arm/Group | GSK2798745
Number analyzed (Participants) | 0

25. Secondary Outcome: Volume of Distribution of GSK2798745
Description: Blood samples were collected at indicated time points for PK parameters including volume of distribution of GSK2798745.
Time Frame: At Day 28
Population: as for outcome 23
Arm/Group | GSK2798745
Number analyzed (Participants) | 0

26. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK2798745
Description: Blood samples were collected at indicated time points for PK parameters including Cmax of GSK2798745.
Time Frame: At Day 28
Population: as for outcome 23
Arm/Group | GSK2798745
Number analyzed (Participants) | 0

27. Secondary Outcome: Area Under Concentration-Time Curve (AUC) Over Dosing Interval of GSK2798745
Description: Blood samples were collected at indicated time points for PK parameters including AUC of GSK2798745.
Time Frame: At Day 28
Population: as for outcome 23
Arm/Group | GSK2798745
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: On treatment AEs, SAEs and non-SAEs were collected from the start of the study treatment until the follow-up (up to Day 56, Week 8).
Description: The results are based on the safety analysis population, which comprised the participants who received at least one dose of study treatment.
Arm/Group | GSK2798745
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2798745 (N=16)
Diabetic retinal oedema (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Feeling abnormal (General disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was early terminated as the study met the prespecified threshold for futility for both SD-OCT and BCVA endpoints of the study based on IA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT04292912/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT04292912/SAP_001.pdf